CLINICAL TRIAL: NCT04584190
Title: Drug Survival of Omalizumab in Chronic Urticaria : a Retrospective Multicentric Study
Brief Title: Real Life Use of Omalizumab in Chronic Urticaria
Acronym: XO-DS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Lyon Civil Hospitals - Lyon Sud Hospital Center (Unknown); Tenon Hospital, Paris (Other); Nantes University Hospital (Other); University Hospital, Grenoble (Other); University Hospital, Rouen (Other); Lille University Hospital (Unknown); University Hospital, Bordeaux (Other); Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0327
Record Dates: First submitted 2020-10-06; First posted 2020-10-12 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Chronic Urticaria
Keywords: Chronic urticaria treated with OMALIZUMAB
MeSH Terms: conditions — Chronic Urticaria

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chronic urticaria affects up to 1% of the population. Chronic urticaria refractory to updosing antihistamines can benefit from OMALIZUMAB, which is an anti-IgE IgG1 monoclonal antibody administrated every 4 weeks subcutaneously which represents a cost of nearly 800€/month excluding nurse fees. Efficacy and good tolerance have already been demonstrated in real-life large cohorts of patients. A 6 months treatment duration is proposed before evaluating the efficacy and discontinuating the treatment in the absence of adequate response. Mean duration of chronic urticaria is 3 to 5 years with high standard deviations. Therefore, optimal duration of treatment with OMALIZUMAB is unknown and discontinuation modalities differ between physicians.

The aim of this study is to evaluate the mean duration between initiation and first discontinuation of OMALIZUMAB in patients treated for chronic urticaria and explore the different factors influencing this duration and its outcome.

DETAILED DESCRIPTION:
Chronic urticaria affects up to 1% of the population. Rarely, chronic urticaria may be refractory to updosing four-fold antihistamine drugs and then can be improved with subcutaneous OMALIZUMAB. OMALIZUMAB is available for chronic urticaria since 2015. It is an IgG1 monoclonal antibody targeting IgE and administrated every 4 weeks which represent a cost of nearly 800€/month excluding nurse fees. Efficacy and good tolerance have already been demonstrated in real-life large cohorts of patients. A 6 months treatment duration is proposed before evaluating the efficacy and discontinuating the treatment in the absence of adequate response. Mean duration of chronic urticaria is 3 to 5 yearss with high standard deviations. Therefore, optimal duration of treatment with OMALIZUMAB is unknown and discontinuation modalities differ between physicians.

The aim of this study is to evaluate the mean duration between initiation and first discontinuation of OMALIZUMAB in patients treated for chronic urticaria and explore the different factors influencing this duration and its outcome.

To accomplish this, the investigators will conduct a restrospective analyse of all patients treated with OMALIZUMAB for chronic urticaria from 2010 to 2020 in the major French hospital reference centers for chronic urticaria management : Paris, Lyon, Grenoble, Lille, Bordeaux, Nantes, Rouen, Saint-Etienne, Montpellier.

ELIGIBILITY:
Inclusion criteria:

* chronic spontaneous or inducible urticaria
* treated with omalizumab
* at least once between January the 1st 2010 and july 2020.

Exclusion criteria:

* unknown intiation and discontinuation date of omalizumab
* omalizumab initiated for asthma
* other diagnosis (vascularitis, aquagenic pruritus)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: French referal hospital centers of chronic urticaria managment
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
duration between initiation and first discontinuation of OMALIZUMAB | 1 day
  assessed at the time of inclusion Description: duration between initiation and first discontinuation of OMALIZUMAB

SECONDARY OUTCOMES:
predictive factors of duration between initiation and first discontinuation of omalizumab | 1 day
  predictive factors of duration between initiation and first discontinuation of omalizumab
efficacy of omalizumab and relapse at discontinuation | 1 day
  efficacy of omalizumab and relapse at discontinuation
discontinuation cause | 1 day
  discontinuation cause
rechallenge with omalizumab and efficacy | 1 day
  rechallenge with omalizumab and efficacy
persistance of antihistamine intake at 1year, 2 years and 3 years | at 1year, 2years and 3years
  persistance of antihistamine intake at 1year, 2 years and 3 years
mid and long-term tolerance of omalizumab. | 1 day
  mid and long-term tolerance of omalizumab.

CONTACTS AND LOCATIONS:
Overall Officials: Aurélie Du Thanh, MD, PhD, Principal Investigator — University Hospitals of Montpellier
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC